CLINICAL TRIAL: NCT03394742
Title: Effectiveness of Peer Support on Quality of Life in Recently Diagnosed Breast Cancer Patients - a Randomized Trial
Brief Title: Effectiveness of Peer Support on Quality of Life in Recently Diagnosed Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jyvaskyla (Other)
Collaborators: Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Anu Toija, Doctoral student, University of Jyvaskyla
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Effectiveness of peer support
Record Dates: First submitted 2017-12-20; First posted 2018-01-09 (Actual); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Breast Cancer
Keywords: Peer Group; Quality of Life
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Peer support group received, in addition to usual care, peer support via telephone 1-5 times according to their own preference. Peer support was started at the time between diagnosis and the beginning of treatments.
  Interventions: Behavioral: Peer support
- Control group (No Intervention): The control group received usual care only. For ethical reasons, participants in the control group were not discouraged from seeking peer support by themselves if they felt a need for it.

INTERVENTIONS:
Behavioral: Peer support — Peer support persons are breast cancer survivors, who were educated to give peer support. They contacted participants by telephone.
  Arms: Intervention group

SUMMARY:
This study examines effectiveness of peer support of breast cancer patients. Half of the participants received peer support via telephone in addition to usual care and another half are give the usual care only.

DETAILED DESCRIPTION:
Seriously sick people need social support to maintain their quality of life. Social support may be given by peers, who have experienced the same.

In this study voluntary participants with recently diagnosed breast cancer were randomly allocated to intervention (N=130) or control (N=130) group. The intervention group received, in addition to usual care, peer support via telephone 1-5 times according to their own preference. The control group received usual care only. Peer support was given by volunteered breast cancer survivors who were educated for giving peer support.

ELIGIBILITY:
Inclusion Criteria:

* recently diagnosed primary breast cancer
* no other serious illnesses
* ability to communicate in Finnish or Swedish (official languages in Finland)
* ability to fill in the questionnaires

Exclusion Criteria:

* some other serious illnesses
* inability to communicate in Finnish or Swedish (official languages in Finland)
* inability to fill in the questionnaires

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Participants were women who had breast cancer.
Enrollment: 260 (Actual)
Dates: Start 2014-05-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
A change of health-related quality of life (HRQoL). | From baseline to 3, 6 and 12 months later.
  HRQoL was assessed with a generic 15D instrument.
A change of health-related quality of life (HRQoL). | From baseline to 3, 6 and 12 months later.
  HRQoL was assessed with a disease-specific instrument EORTC QLQ-30 and its breast cancer specific module BR23.

SECONDARY OUTCOMES:
Satisfaction for life | Baseline and 3, 6 and 12 months later.
  Satisfaction for life was assessed with a questionnaire created for this study.
The use of health care services | Baseline and 3, 6 and 12 months later.
  The use of health care services was assessed with a questionnaire create for this study.

CONTACTS AND LOCATIONS:
Overall Officials: Anu Toija, MHS, Principal Investigator — University of Jyvaskyla
Locations (1):
- Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No